CLINICAL TRIAL: NCT04881604
Title: Compressive Therapy by Adjustable Compression Garment (Ready Wrap®) in Breast Cancer-related Lymphedema: Randomized Clinical Trial
Brief Title: Adjustable Compression Wrap Versus Compression Sleeve to Control Breast Cancer-related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Anke Bergmann, phD, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stage 2 compression therapy
Record Dates: First submitted 2021-04-28; First posted 2021-05-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer Related Lymphedema; Lymphedema, Secondary; Lymphedema of Upper Arm; Breast Neoplasms
Keywords: breast cancer lymphedema; compression bandages
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Neoplasm Metastasis; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization will be by lot when the patient enters the study. Envelopes will be made available that will contain a code that determines the allocation of patients in the intervention group experimental or standard.
Who Masked: Outcomes Assessor
Masking Description: Due to the characteristics of the study, it will be blind only to the researcher responsible for analyzing the collected data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Adjustable Compression Wrap (Experimental): Daily use of the adjustable compression wrap on the upper limb with breast cancer-related lymphedema during phase 2 of compressive therapy.
  Interventions: Device: Adjustable Compression Wrap
- Compression Sleeve (Active Comparator): Daily use of the compressive sleeve on the upper limb with breast cancer-related lymphedema during phase 2 of compressive therapy
  Interventions: Device: Compression Sleeve

INTERVENTIONS:
Device: Adjustable Compression Wrap — Delivery, adaptation and guidance for daily use of the Adjustable Compression Wrap. (Ready Wrap® allows for easy use because to be pre-molded system in inelastic material with self-adjusting compressible components according to the size and shape of the upper limb. Due to its compressive properties, it can be used as therapy to control lymphedema. The material composition is: 61% Nylon, 33% Polyurethane, 6% Elastane (Spandex)).
  The institutional protocol for the lymphedema control phase will be respected, in which the orthosis is used at home for the longest possible period, with only removal for bathing and sleeping; furthermore, skin care and therapeutic exercises for the upper limbs must be performed daily.
  Arms: Adjustable Compression Wrap
Device: Compression Sleeve — Delivery, adaptation and guidance for daily use of the Compression sleeve. (Compression Sleeve is a mesh in the shape of a glove that provides compression on the fabrics needed to help control the volume of the limbs. Traditionally used for stage 2 of compressive therapy. The composition of the material is: 64% Nylon, 36% Elastane (Spandex) ).
  The institutional protocol for the lymphedema control phase will be respected, in which the orthosis is used at home for the longest possible period, with only removal for bathing and sleeping; furthermore, skin care and therapeutic exercises for the upper limbs must be performed daily.
  Other Names: Compressive Mesh
  Arms: Compression Sleeve

SUMMARY:
This is a randomized clinical trial, in which the use of an Adjustable compression wrap as a compressive therapy to control the upper limb volume of with lymphedema women secondary to breast cancer will be investigated, in comparison to the use of a compression sleeve conventionally used. It is expected that Adjustable compression wrap will be more effective than standard treatment for the control of lymphedema, in addition to promoting a better quality of life and functionality for women.

DETAILED DESCRIPTION:
This is a randomized clinical trial of medical devices in pivotal stage, simple blind, which aims to evaluate the effectiveness of the use of adjustable compression wrap in controlling the volume of the upper limb of women with lymphedema secondary to breast cancer. It will be carried out in a reference hospital in the treatment of breast cancer in Brazil, with inclusion scheduled for June 2021 and follow-up of up to 1 year.

All volunteers must have stabilized lymphedema in the upper limb secondary to breast cancer and, therefore indicated phase 2 of compressive therapy. According to the sample calculation will be needed72 women to be randomly randomized in a 1: 1 ratio between the experimental intervention group (n = 36) and the standard intervention group (n = 36).

The Intervention consists of compressive therapy in the control phase for lymphedema secondary to breast cancer, in which the Experimental Intervention Group will receive a Adjustable compression wrap (Read Wrap®) while the Standard Intervention Group will receive a standard compressive sleeve for use in the upper limb with lymphedema, according to the institutional routine. The institutional protocol for the lymphedema control phase will be respected, in which the orthosis is used at home for the longest possible period, with only removal for bathing and sleeping; furthermore, skin care and therapeutic exercises for the upper limbs must be performed daily. One guidance booklet and home exercises of the institutional routine will be delivered . During the initial 30 days of treatment, all study participants will be able to be accompanied by a telephone channel that will be provided for questions, guidance and communications of adverse events, in addition to a therapeutic diary that will be delivered at the first appointment and collected after this period, designed to notify relevant information that they consider about the use of compressive therapy such as facilities, difficulties and time of use, symptoms related to the arm and adverse effects that may arise, and to monitor adherence to exercises.

The suspension of treatment before the anticipated end of therapy will occur when adverse effects are observed, such as an increase in the volume of the limb greater than 10% of the last measurement, signs of dermatitis, skin infections or allergy. The case will be evaluated by the physiotherapy team and, when necessary, by the medical team and the necessary procedures will be adopted.

Data collection will take place through the analysis of physical and electronic medical records, interviews and physical examination. The interviews will consist of questionnaires produced by the researchers, in addition to validated questionnaires for the brazilian population. The evaluations will take place in the outpatient clinic of the physiotherapy service of the hospital on the 1st and 30th day of the intervention for immediate evaluation, and will be followed up until 1 years later, to verify the long-term outcome measures.

The analysis of the data will be descriptive and comparative of the intervention groups, in relation to the selected variables and the main outcomes, through the analysis of measures of central tendency, dispersion and frequency distribution. Outcome assessment will be performed by intention to treat, using linear and logistic regression, simple and multiple. For all analyzes the 95% confidence interval will be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Women

1. Age over 18 years
2. Undergo surgical treatment for breast cancer
3. Diagnosed with lymphedema in the upper limb stabilized for a period ≥6 months
4. Indicated the second phase of compressive therapy / treatment of lymphedema

Exclusion Criteria:

1. Women with:

1. Bilateral lymphedema;
2. Lymphedema since the preoperative period;
3. Presence of phlogistic signs in the limb with lymphedema;
4. Treatment of lymphedema (phase 1) in the last three months;
5. Previous history of allergic reaction to the material used for compressive therapy;
6. Active regional or remote disease;
7. In chemotherapy or radiation therapy;
8. Functional changes in the upper limbs prior to the diagnosis of breast cancer;
9. Heart disease and decompensated systemic arterial hypertension; psychiatric, mental, neurological disorders or cognitive deficits that make it impossible to answer the questionnaires.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Arm volume | Assessment of arm volume will be on the before (1st day), 30 days, 6 months and 1 year after enrollment.
  The main outcome is the change in the volume of the upper limb with lymphedema, which will be assessed through the perimeter of the circumference of the limb, and indirectly estimated the volume of the limb using the cone trunk formula.

SECONDARY OUTCOMES:
Tissue characteristics (fibrosis) of the upper limb with lymphedema | The evaluation of the tissue characteristics of the arm will be before (1st day), 30 days, 6 months and 1 year after enrollment.
  Ultrasonography is used, a non-invasive method of capturing images of tissues through the emission of ultrasonic waves, through the evaluation of images obtained by the portable device, it will be possible to characterize the alteration of the dermoepidermal complex and the tissue. subcutaneous tissue of the upper limb with lymphedema. The report will be provided by a professional with experience in using the kinesiological ultrasound method.
Tissue temperature of the upper limb with lymphedema | The tissue temperature of the arm will be before (1st day), 30 days, 6 months and 1 year after enrollment.
  The tempertature of the arm will be assessed by means of thermography. Thermography is a safe, non-invasive imaging method that determines the distribution of body surface temperatures according to the physiological and pathological condition of the tissues. Inflammation, metabolic changes in the subcutaneous tissue and changes in blood supply result in changes in the temperature gradient of the affected area. In this way, the different stages of lymphedema will be related to different patterns of temperature distribution. The body surface temperatures will be recorded by means of a thermal camera and will be taken in the orthostatic position, from the anterior and posterior portions of the limb, at a distance of 2m. Later, these thermometric images will be analyzed using proprietary software. The standard measurement used will be in degrees celsius (ºC).
Health-related quality of life | The evaluation of the Health-related quality of life will be before (1st day), 30 days, 6 months and 1 year after enrollment.
  Health-related quality of life will be assessed using 'European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30' (EORTC QLQ-C30). It is an instrument validated for our population, which scores from 0 to 100, the higher the value the better the quality of life will be.
Upper limb functionality | The evaluation of the Upper limb functionality will be before (1st day), 30 days, 6 months and 1 year after enrollment.
  The functionality of the upper limbs will be assessed by the 'Disabilities of the Arm, Shoulder and Hand Questionnaire' (DASH). It is a validated instrument for our population, consisting of 30 questions that assess the ability to perform certain activities in the last week, regardless of the upper limb used. The score ranges from 0 to 100, the higher the worse the functionality.
Handgrip strength | The handgrip strength assessment will be before (1st day), 30 days, 6 months and 1 year after enrollment.
  Hand grip strength will be assessed by the dynamometer for 3 attempts, being considered the best of the 3.

OTHER OUTCOMES:
Adverse effects of treatment | Daily documents during the first 30 days of the intervention. And at 6 and 12 months follow-up.
  Punctuated by self-report and professional inspection.
Treatment costs | Total cost of each therapy within 12 months of follow-up.
  Expenses with material, professional, travel and food for each participant will be researched and noted on a form for later analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Bergmann, PhD, Principal Investigator — National Cancer Institute (INCA-BRAZIL)
Locations (1):
- Anke Bergmann, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva JMP, Araujo RDD, da Silva Santos FC, Fabro EAN, de Mello Pinto MV, de Aguiar SS, Thuler LCS, Bergmann A. Complex physical therapy employing self-adjusting garment (ReadyWrap(R)) in breast cancer-related lymphedema cases in Brazilian women: a protocol for a randomized controlled trial. Trials. 2023 Aug 22;24(1):549. doi: 10.1186/s13063-023-07460-4. PMID 37608354